CLINICAL TRIAL: NCT01362153
Title: An Open-label Randomized Phase 1 Study to Investigate the Pharmacokinetics and Pharmacodynamics of Subcutaneous and Intravenous Administrations of Golimumab to Subjects With Rheumatoid Arthritis
Brief Title: A Pharmacokinetic (PK) and Pharmacodynamic (PD) Study of Golimumab in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015550; C0524T14 (Other: Centocor)
Record Dates: First submitted 2011-03-10; First posted 2011-05-30 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Golimumab; Simponi; Rheumatoid Arthritis; PK; PD
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- 001 (Experimental): Golimumab IV infusions of 2 mg/kg golimumab on Days 1 and 85.
  Interventions: Drug: Golimumab
- 002 (Experimental): Golimumab SC injection of 100 mg every 4 weeks through Week 20
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — SC injection of 100 mg every 4 weeks through Week 20
  Arms: 002
Drug: Golimumab — IV infusions of 2 mg/kg golimumab on Days 1 and 85.
  Arms: 001

SUMMARY:
This is a Phase 1, pharmacokinetic and pharmacodynamic study of intravenous and subcutaneous administered golimumab in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
A Phase 1, randomized (study drug route of administration assigned by chance), open label (both physician and patient know that golimumab has been assigned), study of golimumab in patients with rheumatoid arthritis (RA). The purpose of this study is to compare the pharmacokinetic (how the body effects the drug) and pharmacodynamic (how the drug effects the body) effects of golimumab administered through a vein in the arm or by injection under the skin. Safety assessments will be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (eg, blood pressure), and the occurrence and severity of adverse events. The study will also assess the clinical effects of golimumab on RA. The study is planned for approximately 45 patients, which are randomized at a 2:1 ratio to receive golimumab SC or IV. Male or female patients who have been diagnosed with RA for at least 3 months and who are 18 years of age or older may be able to participate. Subcutaneous (SC) injections of 100 mg golimumab every 4 weeks through Week 20 or intravenous (IV) administrations of 2 mg/kg golimumab on Days 1 and 85.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of RA for at least 3 months prior to screening
* Have no history of latent or active tuberculosis (TB) and test negative for TB

Exclusion Criteria:

* Have inflammatory diseases other than RA
* Have been treated with disease-modifying anti-rheumatic drugs (DMARDs)/systemic immunosuppressives other than methotrexate (MTX), sulfasalazine, or hydroxychloroquine during the 4 weeks prior to the first administration of study agent
* Have received intramuscular (IM), IV, or intra-articular corticosteroids within 4 weeks of study agent administration
* Have a known hypersensitivity to human Ig proteins
* Have received infliximab, golimumab, adalimumab or abatacept within 3 months, or etanercept or anakinra within 1 month prior to the first administration of study agent
* Have received alefacept, efalizumab, natalizumab, rituximab, or any B-cell-depleting agent
* Have been treated with any other biologics or investigational drugs, within 5 half-lives of that drug prior to the first administration of study agent
* Have a history of latent or active granulomatous infection, including tuberculosis (TB), histoplasmosis, or coccidioidomycosis, prior to screening
* Have had a Bacille Calmette-Guerin (BCG) vaccination within 12 months of screening
* Have had a serious infection (eg, hepatitis, pneumonia, pyelonephritis, or sepsis)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-12-26 (Actual); Primary Completion 2009-02-27 (Actual); Study Completion 2009-02-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) (Cmax, AUClast, AUCinf, t1/2, systemic clearance, and volume of distribution) following IV administration | 169 days
Pharmacokinetics (PK) [Cmax, tmax, AUC (0-4wk), t1/2 for last dose only, R[AUC(0-4wk)] following SC administration | 211 days
Plasma concentrations of golimumab following IV administration | 169 days
Plasma concentrations of golimumab following SC administration | 211 days

SECONDARY OUTCOMES:
Pharmacodynamics (PD), including C-reactive protein, IL 6, serum amyloid A, tumor necrosis factor alpha, IL 18, E selectin, vascular endothelial growth factor, matrix metalloproteinases, leptin, and haptoglobin | up to 211 days
ACR (American College of Rheumatology) scores | up to 169 days
The number and severity of adverse events | up to 211 days
Efficacy as assessed by percent change in the American College of Rheumatology (ACR) score | up to 169 days

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (9):
- United States (9):
  - Glendale, Arizona
  - Aventura, Florida
  - Palm Harbor, Florida
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Worcester, Massachusetts
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Houston, Texas

REFERENCES:
- [Derived] Doyle MK, Rahman MU, Frederick B, Birbara CA, de Vries D, Toedter G, Wu X, Chen D, Ranganath VK, Westerman ME, Furst DE. Effects of subcutaneous and intravenous golimumab on inflammatory biomarkers in patients with rheumatoid arthritis: results of a phase 1, randomized, open-label trial. Rheumatology (Oxford). 2013 Jul;52(7):1214-9. doi: 10.1093/rheumatology/kes381. Epub 2013 Feb 14. PMID 23418046
- [Derived] Zhuang Y, Xu Z, Frederick B, de Vries DE, Ford JA, Keen M, Doyle MK, Petty KJ, Davis HM, Zhou H. Golimumab pharmacokinetics after repeated subcutaneous and intravenous administrations in patients with rheumatoid arthritis and the effect of concomitant methotrexate: an open-label, randomized study. Clin Ther. 2012 Jan;34(1):77-90. doi: 10.1016/j.clinthera.2011.11.015. Epub 2011 Dec 14. PMID 22169051
- See also: An Open-label Randomized Phase 1 Study to Investigate the Pharmacokinetics and Pharmacodynamics of Subcutaneous and Intravenous Administrations of Golimumab to Subjects with Rheumatoid Arthritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1&filename=CR015550_CSR.pdf